CLINICAL TRIAL: NCT00756535
Title: Exercise Training in a Geriatric Hospital Ward
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Center of the City of Joensuu (Other)
Responsible Party: Leena Timonen, MD,PhD, Chief physician, Health Center of the City of Joensuu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JOE2008
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Frail Elderly
Keywords: Exercise Therapy; Length of Stay; Disability Evaluation
MeSH Terms: interventions — Exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group-based exercise training during hospitalization
  Interventions: Procedure: Exercise training
- 2 (Active Comparator): Usual treatment and rehabilitation during hospitalization
  Interventions: Procedure: usual treatment and rehabilitation

INTERVENTIONS:
Procedure: Exercise training — Group-based exercise training 5 days a week during hospitalization
  Arms: 1
Procedure: usual treatment and rehabilitation — usual treatment and rehabilitation
  Arms: 2

SUMMARY:
The aim of the study is to describe the effects of physical exercise consisting of strength, balance and flexibility training on functional abilities and the length of stay in older (+75) patients hospitalized in a primary-care health- center hospital.

DETAILED DESCRIPTION:
Hospitalization of older people is connected with several adverse events. Hospitalization increases the risk of disability and long-term institutionalization. Immobilization during hospitalization can lead to deterioration of muscle strength and falls. Earlier studies have shown that strength training is beneficial even in the oldest old. Rehabilitation based on strength training exercises can prevent decline in functional capacity and shorten the length of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* age 75 years or older
* ability to walk independently or assisted or move unassisted in a wheelchair

Exclusion Criteria:

* patients in long-term care
* those who are bedridden
* severe circulatory disease
* acute bone fracture
* terminal disease
* acute infection.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Changes in functional abilities during hospitalization | at the discharge from the hospital

SECONDARY OUTCOMES:
The length of stay in the hospital | at the discharge from the hospital

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Health Center of the City of Joensuu, Joensuu, Pohjois-Karjala
  - Siilainen Hospital ward 1A, Joensuu, Pohjois-Karjala

REFERENCES:
- [Background] Rydwik E, Frandin K, Akner G. Effects of physical training on physical performance in institutionalised elderly patients (70+) with multiple diagnoses. Age Ageing. 2004 Jan;33(1):13-23. doi: 10.1093/ageing/afh001. PMID 14870716